CLINICAL TRIAL: NCT00095199
Title: Randomized Phase III Study of Docetaxel or Pemetrexed With or Without Cetuximab in Patients With Recurrent or Progressive Non-Small Cell Lung Cancer After Platinum-Based Therapy
Brief Title: Docetaxel or Pemetrexed With or Without Cetuximab in Patients With Recurrent or Progressive Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13423; I4E-MC-JXBC (Other: Eli Lilly and Company); CP02-0452 (Other: ImClone)
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Recurrent or Progressive Non-Small Cell Lung Cancer; Second-line therapy; Docetaxel; Pemetrexed; Cetuximab; Failed platinum-based therapy; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Pemetrexed; Cetuximab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cetuximab & Pemetrexed (Experimental)
  Interventions: Drug: Pemetrexed; Biological: Cetuximab
- Pemetrexed (Active Comparator)
  Interventions: Drug: Pemetrexed
- Cetuximab & Docetaxel (Experimental)
  Interventions: Biological: Cetuximab; Drug: Docetaxel
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week) cycles.
  Other Names: Alimta; LY231514
  Arms: Cetuximab & Pemetrexed; Pemetrexed
Biological: Cetuximab — Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles until disease progression or unacceptable toxicity.
  Other Names: Erbitux; LY2939777
  Arms: Cetuximab & Docetaxel; Cetuximab & Pemetrexed
Drug: Docetaxel — Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week) cycles.
  Arms: Cetuximab & Docetaxel; Docetaxel

SUMMARY:
This trial is a multicenter, open-label, randomized, Phase III study in patients with recurrent or progressive Non-Small Cell Lung Cancer (NSCLC) after failure of an initial platinum-based chemotherapy. Patients will receive either Docetaxel or Pemetrexed as chemotherapy at the investigator's choice. Within each chemotherapy group, patients will be randomized to receive Cetuximab plus chemotherapy or chemotherapy alone (Cetuximab & Pemetrexed or Pemetrexed alone; Cetuximab & Docetaxel or Docetaxel alone).

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of metastatic, unresectable, or locally-advanced NSCLC.
* Disease progression during or following one prior platinum-based chemotherapy regimen for advanced disease (stage IIIB or IV).
* Bidimensionally measurable disease.
* Karnofsky performance status score of 60 to 100 at study entry.
* The participant has tumor tissue available for immunohistochemical determination of epidermal growth factor (EGFR) expression.
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 4 weeks must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent, or prior radiation therapy (palliative radiation therapy is allowed).
* Accessible for treatment and follow-up. Participants enrolled in this trial must be treated at the participating center.
* Women of childbearing potential (WOCBP) and fertile men with partners of childbearing potential must be using an adequate method of contraception.
* WOCBP must have a negative serum or urine pregnancy test.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* A serious uncontrolled medical disorder that would impair the ability of the patient to receive protocol therapy.
* Symptomatic or uncontrolled metastases in the brain. Participants receiving a glucocorticoid for brain metastases will be excluded, but those receiving anticonvulsants will be eligible.
* Uncontrolled pleural effusion or ascites.
* Peripheral neuropathy greater than grade 2, as assessed by the National Cancer Institutes-Common Toxicity Criteria Adverse Events (NCI-CTCAE), Version 3.0.
* Any concurrent malignancy other than basal cell skin cancer, or carcinoma in situ of the cervix. Patients with a previous malignancy, but without evidence of disease for greater than or equal 3 years will be allowed to enter the trial.
* More than one prior chemotherapy regimen for advanced disease.
* Inadequate hematologic function defined by an absolute neutrophil count (ANC) <1,500/mm3, a platelet count <100,000/mm3, and a hemoglobin level <9 g/dL. Red blood cell transfusions are not permitted within 7 days of receiving cetuximab, docetaxel, or pemetrexed.
* Inadequate hepatic function, defined by a total bilirubin level >1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and alanine aminotransferase (ALT) levels >2.5 times the ULN (greater than or equal to 5 times the ULN if known liver metastases), and an alkaline phosphatase level >5.0 times the ULN.
* Inadequate renal function defined by a serum creatinine level >1.5 times the ULN.
* Prior treatment with cetuximab, or any other epidermal growth factor receptor inhibitors, including tyrosine kinase inhibitors, such as gefitinib or erlotinib. Participants must not have received prior chimerized or murine monoclonal antibody therapy. Prior treatment with other monoclonal antibodies targeting receptors other than the EGFR is permitted >30 days prior to randomization.
* Prior treatment with docetaxel or pemetrexed therapy.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Inability or unwillingness to interrupt nonsteroidal anti-inflammatory drugs (NSAIDs) for a 5-day period (8-day period for long-acting agents such as piroxicam). Aspirin will be permitted during the study.
* Patients (including prisoners) who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Prior treatment with an experimental drug or medical device within 30 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2005-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (67):
- United States (61):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montgomery, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuscon, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stamford, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Worth, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Clemens, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Louis Park, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Joseph, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cary, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., High Point, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hilton Head Island, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mt. Pleasant, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bedford, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grapevine, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colchester, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Jérôme, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec

REFERENCES:
- [Derived] Kim ES, Neubauer M, Cohn A, Schwartzberg L, Garbo L, Caton J, Robert F, Reynolds C, Katz T, Chittoor S, Simms L, Saxman S. Docetaxel or pemetrexed with or without cetuximab in recurrent or progressive non-small-cell lung cancer after platinum-based therapy: a phase 3, open-label, randomised trial. Lancet Oncol. 2013 Dec;14(13):1326-36. doi: 10.1016/S1470-2045(13)70473-X. Epub 2013 Nov 12. PMID 24231627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 939 participants were initially randomized, 1 participant's data was inadvertently lost by a site prior to being entered into the database. As a result, we are reporting 938 as randomized.
Groups:
- Cetuximab & Pemetrexed: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles, until disease progression or unacceptable toxicity. Pemetrexed 500 mg/m^2 administered intravenously on day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week) cycles.
- Pemetrexed: Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 week cycle for up to six (3-week) cycles.
- Cetuximab and Docetaxel: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles until disease progression or unacceptable toxicity. Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
Period: Overall Study
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab and Docetaxel | Docetaxel
Started | 302 (1 participant has no data in database; not included in analyses. Data was lost/destroyed at site.) | 304 | 167 | 166
Completed | 6 | 62 | 7 | 23
Not Completed | 296 | 242 | 160 | 143
Not completed — Adverse Event | 40 | 22 | 26 | 11
Not completed — Progressive disease | 213 | 179 | 105 | 98
Not completed — Death | 10 | 6 | 11 | 9
Not completed — Withdrawal by Subject | 21 | 16 | 13 | 22
Not completed — Protocol Violation | 4 | 4 | 2 | 0
Not completed — Liver function test results elevated | 0 | 0 | 1 | 1
Not completed — Surgery needed could not start in 7 days | 0 | 0 | 1 | 0
Not completed — Physician Decision | 5 | 6 | 1 | 1
Not completed — Not eligible | 1 | 7 | 0 | 1
Not completed — Started Palliative Radiotherapy | 1 | 0 | 0 | 0
Not completed — Started radiotherapy regimen | 0 | 1 | 0 | 0
Not completed — Primary tumor removed in other surgery | 0 | 1 | 0 | 0
Not completed — Data inadvertently lost by site | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cetuximab & Pemetrexed: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles until disease progression or unacceptable toxicity. Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week) cycles.
- Cetuximab & Docetaxel: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles until disease progression or unacceptable toxicity. Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
- Total: Total of all reporting groups
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel | Total
Number analyzed (Participants) | 301 | 304 | 167 | 166 | 938
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.0) | 64.0 (9.4) | 63.6 (9.4) | 63.9 (9.2) | 63.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 116 | 75 | 73 | 392
  Male | 173 | 188 | 92 | 93 | 546
Race/Ethnicity, Customized [Number; unit: participants]
  White | 268 | 265 | 146 | 141 | 820
  Black or African American | 25 | 24 | 13 | 20 | 82
  Asian | 3 | 6 | 5 | 2 | 16
  Hispanic | 4 | 8 | 2 | 2 | 16
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 265 | 270 | 152 | 151 | 838
  Canada | 36 | 34 | 15 | 15 | 100
Epidermal growth factor receptor (EGFR) by immunohistochemistry [Number; unit: participants] — Immunohistochemical staining intensity of anti-EGFR antibody: Score 0=No staining is observed in membrane; Score +1=Staining in membrane is partial, weak and barely perceptible; Score +2=Staining is weak but is completely observed in membrane; Score +3=Strong complete membrane staining is observed. EGFR positive staining is a potential prognostic factor in non-small cell lung cancer. Presence of EGFR staining was not, however, an inclusion criteria or used to stratify participants in the trial.
  participants
    +1 | 36 | 35 | 13 | 19 | 103
    +2 | 46 | 53 | 26 | 34 | 159
    +3 | 118 | 108 | 72 | 58 | 356
    0 | 21 | 32 | 12 | 10 | 75
    Missing | 80 | 76 | 44 | 45 | 245
Karnofsky Performance Status [Number; unit: participants] — Karnofsky performance status was part of eligibility criteria and classifies participants according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses. 100=Normal. No complaints. No evidence of disease; 90=Able to carry on normal activity. Minor signs of disease; 80=Activity with effort. Some signs of disease; 70=Unable to carry on normal activity or to do active work; 60=Requires occasional assistance, but is able to care for most needs; <60=Needs increasing assistance, up to a score of 0=death.
  participants
    60 | 12 | 14 | 2 | 11 | 39
    70 | 35 | 35 | 21 | 14 | 105
    80 | 103 | 91 | 55 | 57 | 306
    90 | 101 | 116 | 74 | 64 | 355
    100 | 48 | 47 | 14 | 18 | 127
    Missing/unknown | 2 | 1 | 1 | 2 | 6
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma | 161 | 185 | 99 | 83 | 528
  Large cell carcinoma | 19 | 7 | 7 | 3 | 36
  All other non-squamous diagnoses | 45 | 41 | 20 | 29 | 135
  Squamous cell carcinoma | 76 | 71 | 41 | 51 | 239

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization until the date of progressive disease (PD) or death from any cause. Participants who were alive and without progression were censored at the date of their last tumor assessment. PFS was assessed by the independent review committee (IRC) in the Pemetrexed group (Cetuximab & Pemetrexed versus Pemetrexed) and by the investigator in the Docetaxel group (Cetuximab & Docetaxel versus Docetaxel).
Time Frame: Randomization to progression of disease or death due to any cause up to 59.6 months
Population: The intent-to-treat population (ITT) included all participants classified according to the treatment arms into which they were randomized, regardless of the actual treatment received. Censored participants: 10 in Cetuximab + Pemetrexed arm; 25 in Pemetrexed arm; 6 in Cetuximab + Docetaxel arm; 16 in Docetaxel arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cetuximab & Pemetrexed: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week) cycles until disease progression or unacceptable toxicity. Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week cycles).
- Pemetrexed: Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
- Cetuximab & Docetaxel: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously every 3 weeks cycle for up to six (3-week) cycles, after 6 cycles participants on the chemotherapy/cetuximab combination may continue cetuximab alone. Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
- Docetaxel: Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 301 | 304 | 167 | 166
months | 2.89 [2.69 to 3.22] | 2.76 [2.53 to 3.29] | 2.37 [1.61 to 2.89] | 1.54 [1.45 to 2.50]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; The Pemetrexed comparisons (Cetuximab + Pemetrexed vs Pemetrexed) were considered the primary comparisons. The Docetaxel comparisons (Cetuximab + Docetaxel vs Docetaxel) were considered supportive as Docetaxel comparisons remained underpowered by design. No tests were conducted to compare participants who received Docetaxel to those who received Pemetrexed; Test type: Superiority or Other; p = 0.756, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; Kaplan-Meier method estimated median PFS time. HR was calculated with unstratified Cox proportional hazards model. HR<1 favours Cetuximab arm; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.87 to 1.21]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.391, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.13]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death. Participants without a date of death were censored on the last date participants were known to be alive, or lost to follow-up.
Time Frame: Randomization to the date of death from any cause up to 72.8 months
Population: The intent-to-treat population (ITT) included all participants classified according to the treatment arms into which they were randomized, regardless of the actual treatment received. Censored participants: 24 in Cetuximab + Pemetrexed arm; 43 in Pemetrexed arm; 12 in Cetuximab + Docetaxel arm; 22 in Docetaxel arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 301 | 304 | 167 | 166
months | 6.93 [6.28 to 7.85] | 7.79 [6.77 to 8.41] | 5.75 [4.73 to 8.31] | 8.15 [6.11 to 9.20]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.864, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; Kaplan-Meier method estimated median OS time. HR was calculated with unstratified Cox proportional hazards model. HR<1 favors Cetuximab arm; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.86 to 1.20]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.307, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.90 to 1.41]

3. Secondary Outcome: Proportion of Randomized Participants With the Best Overall Response (OR) of Partial Response (PR) or Complete Response (CR) (Overall Response Rate [ORR])
Description: The best overall response rate (ORR) was the proportion of randomized participants with a best OR of CR or PR, according to modified World Health Organization (WHO) guidelines. It was calculated as the total number of participants with CR or PR divided by the total number of participants treated in that arm. Participants with no post-baseline evaluation were considered as non-responders. The tumor response was assessed by the independent review committee (IRC) in the Pemetrexed group and by the investigator in the Docetaxel group.
Time Frame: Randomization until progression of disease or death from any cause up to 59.6 months
Population: The intent-to-treat population (ITT) included all participants classified according to the treatment arms into which they were randomized, regardless of the actual treatment received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 301 | 304 | 167 | 166
proportion of participants | 0.066 [0.038 to 0.095] | 0.043 [0.020 to 0.066] | 0.078 [0.037 to 0.118] | 0.066 [0.028 to 0.104]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.200, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.78 to 3.26]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.683, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.52 to 2.74]

4. Secondary Outcome: Proportion of Randomized Participants With Best Overall Response (OR) of Partial Response (PR), Complete Response (CR), or Stable Disease (SD)
Description: The disease control rate (DCR) was the proportion of randomized participants with a best OR of CR, PR or SD according to modified World Health Organization (WHO) guidelines. It was calculated as the total number of participants with CR, PR or SD divided by the total number of participants randomized in that arm. The tumor response was assessed by the independent review committee (IRC) in the Pemetrexed group and by the investigator in the Docetaxel group.
Time Frame: Randomization to progression of disease or death due to any cause up to 59.6 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 301 | 304 | 167 | 166
proportion of participants | 0.522 [0.465 to 0.578] | 0.480 [0.424 to 0.536] | 0.335 [0.264 to 0.407] | 0.253 [0.187 to 0.319]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.310, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.86 to 1.62]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.100, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.93 to 2.40]

5. Secondary Outcome: Percentage of Participants With Symptomatic Response (Symptom Response Rates) Using the Lung Cancer Subscale (LCS) Scores of Functional Assessment of Cancer Therapy for Participants With Lung Cancer (FACT-L)
Description: The FACT-LCS is a set of 7 questions to inventory problems specific to lung cancer symptoms. Participants rate each item on a 5-point Likert-type scale from 0 (not at all) to 4 (very much). Scores range from 0-28 and higher score indicates fewer symptoms. Symptom response (improvement) was defined as ≥2 point increase from baseline in the 7-item LCS score that was maintained for 2 consecutive assessments at least 3 weeks, and not >5 weeks apart for participants, whose baseline LCS score was ≤26. Symptom response rate was the percentage of participants with symptomatic response.
Time Frame: At baseline, every 3 weeks and 30 days after end of therapy up to 50 months
Population: The randomized participants with baseline LCS scores less than or equal to 26.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 280 | 280 | 150 | 155
percentage of participants | 17.1 [12.7 to 21.6] | 22.9 [17.9 to 27.8] | 17.3 [11.3 to 23.4] | 13.5 [8.2 to 18.9]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.091, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.46 to 1.06]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.361, Mantel Haenszel — The 2-sided unstratified Mantel Haenszel test was employed at the 5% significance level; HR<1 favors Cetuximab arm; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.72 to 2.50]

6. Secondary Outcome: Time to Symptomatic Progression
Description: The FACT-LCS (see description in Outcome measure 5) inventories problems specific to lung cancer symptoms. Using this Scale, Symptom progression = a ≥ 2 point decrease from baseline in LCS score maintained for 2 consecutive assessments ≥3 weeks, and <5 weeks, apart. The symptom progression date = the first of 2 consecutive assessments with a ≥2 point decline. Time to symptomatic progression = the time from randomization to the symptom progression date. For participants with no symptom progression, time to symptomatic progression was censored the date of last symptom assessment.
Time Frame: Randomization until symptomatic progression up to 48.3 months
Population: All randomized participants with a baseline LCS >= 2 were included. Censored participants: 237 in Cetuximab plus Pemetrexed arm; 244 in Pemetrexed arm; 126 in Cetuximab plus Docetaxel arm; 131 in Docetaxel arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cetuximab & Docetaxel: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously every 3 weeks cycle for up to six (3-week cycles), after 6 cycles participants on the chemotherapy/cetuximab combination may continue cetuximab alone. Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week) cycles.
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 289 | 287 | 152 | 158
months | NA [NA to NA] — The median time to symptomatic progression is not estimable because the probability of symptomatic progression free never decreased to 0.5 | NA [NA to NA] — The median time to symptomatic progression is not estimable because the probability of symptomatic progression free never decreased to 0.5 | NA [7.00 to NA] — The median time to symptomatic progression is not estimable because the probability of symptomatic progression free never decreased to 0.5 | NA [NA to NA] — The median time to symptomatic progression is not estimable because the probability of symptomatic progression free never decreased to 0.5
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.472, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; Kaplan-Meier estimated time to symptomatic progression. HR was calculated using unstratified Cox proportional hazards model. HR<1 favors Cetuximab arm; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.77 to 1.74]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.272, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; [statistical method as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.42 to 1.27]

7. Secondary Outcome: Duration of Overall Response (OR)
Description: The duration of response, in participants with best OR of complete response (CR) or partial response (PR), was measured from the date criteria are met for CR/PR (not confirmation date, whichever was first recorded), until the first occurrence date that the criteria of progressive disease (PD) was met, or death. Participants who were alive and without progression were censored at the date of their last independent review committee (IRC) tumor assessment. The tumor response and progression were assessed by the IRC in the Pemetrexed group and by the investigator in the Docetaxel group.
Time Frame: Time of first occurrence of either (PR) or (CR) to the first date of progressive disease or death up to 32.5 months
Population: All randomized participants with a best overall response of CR or PR. Censored participants: 1 in Cetuximab plus Pemetrexed arm; 2 in Pemetrexed arm; 1 in Cetuximab plus Docetaxel arm; 0 in Docetaxel arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cetuximab & Docetaxel: Cetuximab 400/250 mg/m2 (initial/weekly) administered intravenously every 3 weeks cycle for up to six (3-week) cycles, after 6 cycles participants on the chemotherapy/cetuximab combination may continue cetuximab alone. Docetaxel 75 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle for up to six (3-week cycles).
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab & Docetaxel | Docetaxel
Number analyzed (Participants) | 20 | 13 | 13 | 11
months | 4.17 [2.92 to 5.45] | 6.93 [3.98 to 16.36] | 5.36 [2.73 to 6.93] | 5.39 [3.12 to 7.16]
Statistical Analysis 1: Comparison: Cetuximab & Pemetrexed vs Pemetrexed; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.236, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; The Kaplan-Meier method estimated duration of response. HR was calculated using unstratified Cox proportional hazards model. HR<1 favors Cetuximab arm; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [0.74 to 3.36]
Statistical Analysis 2: Comparison: Cetuximab & Docetaxel vs Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.887, Log Rank — The 2-sided unstratified log-rank test was employed at the 5% significance level; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.42 to 2.18]

8. Secondary Outcome: Number of Participants With Common Toxicity Criteria (CTC) Grade 3 or 4 Toxicities
Description: National Cancer Institutes-Common Toxicity Criteria version 3.0 was used by investigators to assess participant toxicities. Mapping of investigator verbatim terms to CTCAE terms was done by the sponsor/designee using CTCAE v4.0. Participants reported had grade 3 or 4 toxicities (or both potentially). Grade 3 AEs: severe or medically significant but not immediately life-threatening;hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4 AEs: life-threatening consequences; urgent intervention indicated.
Time Frame: Time from first dose to 30 days after last dose of study therapy up to 28.3 months for Cetuximab & Pemetrexed (versus Pemetrexed alone) and up to 54.3 months for Cetuximab + Docetaxel (versus Docetaxel alone)
Population: All randomized participants receiving at least 1 dose of study drug made up the safety population for this outcome measure. Investigators graded events using CTCAE v3.0. Mapping of investigator verbatim terms for toxicity to CTCAE terms was done by the sponsor/designee using CTCAE v4.0.
Measure: Number; unit: participants
Groups:
- Cetuximab & Pemetrexed: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Days 1, 8, and 15 (3-week cycles) until disease progression or unacceptable toxicity. Pemetrexed 500 mg/m^2 administered intravenously on Day 1 of 3 weeks cycle until disease progression or unacceptable toxicity for up to six (3-week) cycles.
- Cetuximab + Docetaxel: Cetuximab 400/250 mg/m^2 (initial/weekly) administered intravenously on Day 1 of every 3 weeks cycle for up to six (3-week) cycles, after 6 cycles participants on the chemotherapy/cetuximab combination may continue cetuximab alone. Docetaxel 75 mg/m2 administered intravenously on Day 1 of 3 week cycle for up to six (3-week) cycles.
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab + Docetaxel | Docetaxel
Number analyzed (Participants) | 292 | 289 | 159 | 149
participants | 179 | 143 | 112 | 97

ADVERSE EVENTS:
Time Frame: Randomization to 30 days after study therapy up to 72.8 months for Cetuximab & Pemetrexed (versus just Pemetrexed) and up to 64.3 months for Cetuximab + Docetaxel (versus just Docetaxel)
Arm/Group | Cetuximab & Pemetrexed | Pemetrexed | Cetuximab and Docetaxel | Docetaxel
Serious Adverse Events (participants affected / at risk) | 119/292 | 86/289 | 84/159 | 60/149
Other Adverse Events (participants affected / at risk) | 289/292 | 281/289 | 159/159 | 147/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab & Pemetrexed (N=292) | Pemetrexed (N=289) | Cetuximab and Docetaxel (N=159) | Docetaxel (N=149)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 6 (7) | 2 (2) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 13 (14) | 11 (11)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 10 (11) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (12) | 2 (2) | 0 (0) | 5 (7)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (3) | 1 (1) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (4) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 6 (7) | 1 (1)
Asthenia (General disorders) | 6 (6) | 1 (1) | 4 (4) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 6 (6) | 2 (2) | 5 (5) | 5 (5)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Pain (General disorders) | 5 (5) | 4 (4) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 5 (5) | 10 (10) | 3 (3)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 16 (16) | 17 (17) | 9 (11) | 10 (10)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 11 (11) | 6 (7) | 17 (19) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 6 (6) | 4 (5) | 5 (5) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (5) | 1 (1) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 11 (14) | 12 (13) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3) | 7 (7) | 3 (3)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 4 (5) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 3 (3) | 4 (4) | 7 (10)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (3) | 7 (8) | 3 (6)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain management (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 5 (6) | 0 (0) | 8 (8) | 2 (2)
Exsanguination (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 0 (0) | 5 (6) | 5 (5)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab & Pemetrexed (N=292) | Pemetrexed (N=289) | Cetuximab and Docetaxel (N=159) | Docetaxel (N=149)
Anaemia (Blood and lymphatic system disorders) | 70 (90) | 64 (93) | 40 (75) | 35 (48)
Leukopenia (Blood and lymphatic system disorders) | 10 (14) | 11 (17) | 15 (31) | 7 (13)
Neutropenia (Blood and lymphatic system disorders) | 32 (51) | 32 (58) | 74 (121) | 46 (95)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (26) | 22 (48) | 7 (11) | 2 (7)
Tachycardia (Cardiac disorders) | 13 (16) | 12 (12) | 15 (15) | 8 (8)
Lacrimation increased (Eye disorders) | 20 (21) | 16 (16) | 7 (7) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 19 (22) | 16 (19) | 15 (16) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 16 (18) | 10 (10) | 4 (9) | 3 (3)
Constipation (Gastrointestinal disorders) | 75 (94) | 60 (66) | 41 (48) | 25 (27)
Diarrhoea (Gastrointestinal disorders) | 81 (108) | 36 (38) | 63 (91) | 22 (28)
Dyspepsia (Gastrointestinal disorders) | 21 (26) | 15 (16) | 12 (16) | 7 (7)
Nausea (Gastrointestinal disorders) | 112 (146) | 89 (128) | 53 (68) | 38 (48)
Oral pain (Gastrointestinal disorders) | 11 (12) | 7 (7) | 8 (8) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 54 (78) | 21 (21) | 53 (74) | 23 (26)
Vomiting (Gastrointestinal disorders) | 59 (83) | 44 (54) | 25 (32) | 19 (22)
Asthenia (General disorders) | 37 (40) | 33 (42) | 29 (41) | 15 (20)
Chills (General disorders) | 12 (14) | 13 (13) | 9 (12) | 15 (16)
Fatigue (General disorders) | 158 (209) | 133 (191) | 88 (146) | 74 (99)
Non-cardiac chest pain (General disorders) | 14 (14) | 18 (22) | 6 (7) | 7 (9)
Oedema peripheral (General disorders) | 51 (70) | 32 (35) | 23 (28) | 27 (28)
Pain (General disorders) | 12 (20) | 14 (15) | 10 (12) | 11 (12)
Pyrexia (General disorders) | 46 (60) | 37 (43) | 22 (29) | 14 (14)
Candidiasis (Infections and infestations) | 11 (13) | 5 (6) | 8 (9) | 6 (6)
Oral candidiasis (Infections and infestations) | 9 (11) | 6 (6) | 10 (13) | 5 (7)
Paronychia (Infections and infestations) | 15 (21) | 0 (0) | 3 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 18 (20) | 9 (10) | 8 (9) | 6 (7)
Infusion related reaction (Injury, poisoning and procedural complications) | 15 (19) | 0 (0) | 4 (5) | 2 (2)
Weight decreased (Investigations) | 19 (25) | 15 (15) | 18 (20) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 86 (102) | 58 (63) | 54 (68) | 45 (47)
Dehydration (Metabolism and nutrition disorders) | 27 (28) | 17 (21) | 24 (28) | 14 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (14) | 20 (28) | 6 (7) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 29 (33) | 11 (12) | 26 (32) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 57 (91) | 17 (20) | 36 (55) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (18) | 22 (23) | 14 (18) | 17 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (44) | 14 (16) | 17 (19) | 7 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (12) | 1 (1) | 9 (12) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (12) | 10 (10) | 10 (11) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 (22) | 13 (13) | 7 (9) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 13 (14) | 8 (9) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (25) | 11 (11) | 21 (23) | 14 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (25) | 16 (16) | 11 (14) | 6 (6)
Dizziness (Nervous system disorders) | 41 (49) | 14 (18) | 21 (26) | 18 (22)
Dysgeusia (Nervous system disorders) | 25 (25) | 12 (12) | 23 (30) | 13 (13)
Headache (Nervous system disorders) | 20 (28) | 21 (22) | 8 (8) | 15 (16)
Neuropathy peripheral (Nervous system disorders) | 14 (14) | 15 (15) | 16 (18) | 13 (15)
Anxiety (Psychiatric disorders) | 20 (22) | 16 (18) | 8 (8) | 6 (6)
Confusional state (Psychiatric disorders) | 17 (21) | 13 (15) | 7 (7) | 7 (7)
Depression (Psychiatric disorders) | 16 (17) | 20 (20) | 8 (9) | 9 (9)
Insomnia (Psychiatric disorders) | 27 (29) | 27 (27) | 11 (12) | 19 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (50) | 43 (46) | 28 (31) | 23 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 5 (5) | 5 (7) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 66 (84) | 60 (71) | 43 (61) | 38 (43)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 11 (13) | 19 (21) | 5 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 9 (9) | 10 (15) | 8 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (8) | 8 (9) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 13 (15) | 12 (14) | 11 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 9 (11) | 8 (9) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (20) | 5 (5) | 29 (32) | 36 (36)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 223 (444) | 5 (5) | 100 (160) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 62 (70) | 8 (8) | 27 (34) | 7 (7)
Erythema (Skin and subcutaneous tissue disorders) | 12 (13) | 3 (3) | 9 (12) | 7 (7)
Nail disorder (Skin and subcutaneous tissue disorders) | 17 (20) | 0 (0) | 8 (8) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 30 (36) | 6 (7) | 13 (16) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 20 (35) | 32 (38) | 8 (10) | 12 (13)
Skin disorder (Skin and subcutaneous tissue disorders) | 24 (33) | 0 (0) | 13 (17) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 15 (22) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 29 (34) | 9 (9) | 15 (17) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days